CLINICAL TRIAL: NCT02758119
Title: Conciliating Mastery Learning and Time Constraints on High-fidelity Simulators: Serious Game Versus Online Course to Pre-train Medical Students on the Management of an Adult Cardiac Arrest.
Brief Title: Serious Game Versus Online Course to Pre-train Medical Students on the Management of an Adult Cardiac Arrest.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilumens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ilumens0002
Record Dates: First submitted 2016-04-29; First posted 2016-05-02 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-03

CONDITIONS: Education, Medical, Undergraduate; Out-of-Hospital Cardiac Arrest; Simulation Training
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Serious Game (Experimental): Participants in the "serious game" group will be pre-trained before the hands-on sessions with the serious game "Staying Alive", available at http://www.stayingalive.fr/index_us.html This game aims at teaching the management of an out-of-hospital cardiac arrest to the general public and health professionals. In this game, the player faces a man who has experienced sudden cardiac arrest and learns the appropriate behavior, movements and techniques that can contribute to saving his life. The first level of the game lasts 4-5 minutes, depending on the skills of the player. It is a point and click game, displayed on a PC computer.
  Interventions: Other: Serious Game
- Online course (Active Comparator): Participants in the lecture group will watch individually a 4-min video of a PowerPoint presentation with voiceover narration, given in the medical school of Paris Descartes University. The video is edited to contain the same informations on out-of-hospital cardiac management than the serious game, with the same duration.
  Interventions: Other: Online course

INTERVENTIONS:
Other: Serious Game
  Arms: Serious Game
Other: Online course
  Arms: Online course

SUMMARY:
The objective of this study is to compare two forms of pre-training (an online narrative presentation and a serious game) to prepare 2nd year medical students for a hands-on training with physical simulators about out-of-hospital cardiac arrest management.

DETAILED DESCRIPTION:
Technology-enhanced simulation allows mastery learning. Mastery learning is a variety of competency-based education which has demonstrated its efficacy for skills acquisition and their transfer to actual settings. While traditional education defines fixed learning time and allows outcomes to vary, in mastery learning, all trainees must achieve a predefined level of proficiency while their learning time can vary. The main limitation of mastery learning is that it takes more time than non-mastery learning. This is of concern because the main barrier to simulation-based training is the lack of faculty time. Thus, new solutions should emerge to conciliate mastery learning and time constraints on physical simulators.

Pre-training with a "simulation game" may be a mean to reach this objective. Simulation games are serious games which are at the cross roads between (1) educational games which are "applications using the characteristics of video and computer games to create engaging and immersive learning experiences", and (2) simulation, the imitation of situations which can be encountered in real-life. They combine the advantages of educational games (active, personalized learning) and simulation (realistic and safe environment for experiential learning). By contrast, pre-training with an online course using a PowerPoint presentation with voiceover narration lecture is both passive and abstract.

The objective of this study is to evaluate the time-efficiency of pre-training using a simulation game versus an online course to reach mastery learning in the management of an adult out-of-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Second-year medical students from the medical schools of Paris Descartes and Paris Diderot University who are not opposed to participate in the study.

Exclusion Criteria:

* Opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Drummond, MD, Principal Investigator — University Paris René Descartes
Locations (1):
- Département de Simulation iLumens, Université Paris Descartes, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mundell WC, Kennedy CC, Szostek JH, Cook DA. Simulation technology for resuscitation training: a systematic review and meta-analysis. Resuscitation. 2013 Sep;84(9):1174-83. doi: 10.1016/j.resuscitation.2013.04.016. Epub 2013 Apr 23. PMID 23624247
- [Background] Wayne DB, Butter J, Siddall VJ, Fudala MJ, Wade LD, Feinglass J, McGaghie WC. Mastery learning of advanced cardiac life support skills by internal medicine residents using simulation technology and deliberate practice. J Gen Intern Med. 2006 Mar;21(3):251-6. doi: 10.1111/j.1525-1497.2006.00341.x. PMID 16637824
- [Background] Cook DA, Brydges R, Zendejas B, Hamstra SJ, Hatala R. Mastery learning for health professionals using technology-enhanced simulation: a systematic review and meta-analysis. Acad Med. 2013 Aug;88(8):1178-86. doi: 10.1097/ACM.0b013e31829a365d. PMID 23807104
- [Background] Creutzfeldt J, Hedman L, Fellander-Tsai L. Effects of pre-training using serious game technology on CPR performance--an exploratory quasi-experimental transfer study. Scand J Trauma Resusc Emerg Med. 2012 Dec 6;20:79. doi: 10.1186/1757-7241-20-79. PMID 23217084
- [Derived] Drummond D, Delval P, Abdenouri S, Truchot J, Ceccaldi PF, Plaisance P, Hadchouel A, Tesniere A. Serious game versus online course for pretraining medical students before a simulation-based mastery learning course on cardiopulmonary resuscitation: A randomised controlled study. Eur J Anaesthesiol. 2017 Dec;34(12):836-844. doi: 10.1097/EJA.0000000000000675. PMID 28731928
- See also: Official website of the departement of simulation in healthcare, Paris Descartes University — http://ilumens.fr

RESULTS

PARTICIPANT FLOW:
Groups:
- Online Course: Participants in the lecture group will watch individually a 4-min video of a PowerPoint presentation with voiceover narration, given in the medical school of Paris Descartes University. The video is edited to contain the same informations on out-of-hospital cardiac management than the serious game, with the same duration.
  Online course
- Serious Game: Participants in the "serious game" group will be pre-trained before the hands-on sessions with the serious game "Staying Alive", available at http://www.stayingalive.fr/index_us.html This game aims at teaching the management of an out-of-hospital cardiac arrest to the general public and health professionals. In this game, the player faces a man who has experienced sudden cardiac arrest and learns the appropriate behavior, movements and techniques that can contribute to saving his life. The first level of the game lasts 4-5 minutes, depending on the skills of the player. It is a point and click game, displayed on a PC computer.
  Serious Game
Period: Overall Study
Arm/Group | Online Course | Serious Game
Started | 41 | 41
Completed | 39 | 40
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Serious Game | Online Course | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21 [20 to 21] | 21 [21 to 21] | 21 [21 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Last basic life support course taken, [Count of Participants; unit: Participants]
  Never | 12 | 20 | 32
  < 12 months | 4 | 5 | 9
  > 12 months | 25 | 16 | 41
Familiar with low-fidelity simulation [Count of Participants; unit: Participants] | 11 | 12 | 23
Familiar with high-fidelity simulation [Count of Participants; unit: Participants] | 1 | 0 | 1
Previous participation in CPA management [Count of Participants; unit: Participants] | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Training Time Needed to Reach the Minimal Passing Score for a Simulated Out-of-hospital Cardiac Arrest Scenario Using a High-fidelity Simulator at Day 8.
Description: Following the 2015 European Resuscitation Council guidelines, a checklist was developed for this study. This checklist allows the assessors to evaluate the participant's compliance with guidelines, and to determine if he/she needs to practice again on the scenario or if he/she reached the minimum passing score and can stop the training.
  The quality of the chest compressions provided is recorded automatically through the ResusciAnne Skill Reporter Software (Laerdal, Norways), and is integrated in the checklist.
Time Frame: The hands-on session takes place 8 days after the first pre-training when the serious game or the online course are played/watched twice, and one day after the second pre-training when they are played/watched once more
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Online Course | Serious Game
Number analyzed (Participants) | 39 | 40
minutes | 23 [15 to 32] | 20.5 [15.8 to 30.3]

2. Secondary Outcome: Median Training Time Needed to Reach the Minimal Passing Score for a Simulated Out-of-hospital Cardiac Arrest Scenario Using a High-fidelity Simulator
Description: Evaluation of skill retention.
Time Frame: 4 months after the hands-on session.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Serious Game | Online Course
Number analyzed (Participants) | 38 | 37
Minutes | 11.7 [10.7 to 17.0] | 12.1 [10.2 to 21.5]
Statistical Analysis 1: Comparison: Serious Game vs Online Course; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Score (on the Checklist) on the First Attempt During the hands-on Session
Description: Name: Checklist for performance score of SCA management This checklist was adapted from the 2015 resuscitation guidelines. Points were given for the actions performed correctly in sequence and in time(sequence score, 0 to 4),and for the quality of the chest compressions (compression score,0 to 8). The minimum passing score on this checklist was 11 out of 12 (min 0-max 12), with the absolute requirement to score the maximum 4 points on the sequence score.
  Higher scores mean a better outcome.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Serious Game | Online Course
Number analyzed (Participants) | 40 | 39
units on a scale | 6 [4 to 8] | 6 [5 to 7]

4. Secondary Outcome: Score (on the Checklist) on the First Attempt During the hands-on Session
Description: as for outcome 3
Time Frame: 4 months after the hands-on session.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Serious Game | Online Course
Number analyzed (Participants) | 38 | 37
units on a scale | 9 [8 to 10] | 9 [8 to 10]

ADVERSE EVENTS:
Arm/Group | Online Course | Serious Game
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No